CLINICAL TRIAL: NCT01056458
Title: Effect of Auricular Acupressure on Perimenopausal and Early Postmenopausal Women With Anxiety: a Double Blinded, Randomized and Controlled Study
Brief Title: Auricular Acupressure for Perimenopausal Women With Anxiety
Acronym: AAA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang-Hua Hospital (Other Government)
Collaborators: China Medical University Hospital (Other)
Responsible Party: Ching-Ling Kao, MD, Chang-Hua Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 98DMR291
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2010-05-31 (Estimated); Status verified 2010-01

CONDITIONS: Auricular Acupressure; Anxiety; Menopause; Insomnia
Keywords: acupressure; perimenopause; menopause; anxiety; life quality; insomnia
MeSH Terms: conditions — Anxiety Disorders; Sleep Initiation and Maintenance Disorders | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupressure acupressure (Active Comparator)
  Interventions: Other: auricular acupressure
- sham acupressure (Sham Comparator)
  Interventions: Other: sham acupressure

INTERVENTIONS:
Other: auricular acupressure — use the tape of ear adhesive beads on shenmen and subcortical area of both ears after three meals and before bed for three minutes each area with alternating ears, twice a week to replace paste.
  Other Names: acupressure
  Arms: Acupressure acupressure
Other: sham acupressure — use only tape without ear adhesive beads under the same ways
  Other Names: acupressure
  Arms: sham acupressure

SUMMARY:
This study is expected to show auricular acupressure therapy help to improve the anxiety symptoms of perimenopausal and early postmenopausal women, looking forward to developing a convenient, safe and effective way to reduce the use of sedative hypnotics and their dependencies, thereby improving their quality of life.

DETAILED DESCRIPTION:
There are several stages of women while they were particularly vulnerable to anxiety and insomnia , especially in the pre-menstruation, pregnancy, postpartum, and menopause stage. Sleep problems are common in menopausal and postmenopausal women, its prevalence can be based on research from 15% to 60%. As for anxiety, the prevalence of women in this population can reach 53.7%. Several studies overseas have already pointed out that the improvement of acupuncture for anxiety disorders have had pretty good results. As auricular acupressure with a simple operation and the advantages of non-invasive, our interest is to explore the clinical benefit of combined auricular acupressure and medical therapy on anxiety and insomnia improvement in menopausal and early post-menopausal women. We design a double-blind, randomized controlled study, the subjects are ninety 40 to 60 years old women, during perimenopause and early postmenopause who are accompanied by anxiety symptoms. They were randomly divided into experimental and control groups, use the tape of ear adhesive beads on shenmen and subcortical area of both ears after three meals and before bed for three minutes each area with alternating ears, twice a week to replace paste. A total treatment time is eight times and a total of four weeks. Primary efficacy assessment (primary outcome measure) for the Hamilton Anxiety Rating Scale (HAMA) total score change. Secondary efficacy assessments (secondary outcome measure) for: 1) Menopause Rating Scale (MRS) scores; 2) Short Form Health Survey (SF-36) scores; 3) Clinical Global Impression-Severity (CGI-S) scores; and 4) Clinical Global Impression-Improvement (CGI-I) score changes.

ELIGIBILITY:
Inclusion Criteria:

* age between 40 to 60 years
* irregular menstrual cycle less than 12 months or no menstrual cycle less than 10 years
* FSH level>= 14 IU/L
* Brief symptom rating scale total scores>= 6

Exclusion Criteria:

* severe medical conditions
* substance dependence or abuse
* contraindication of BZDs
* contraindication of acupressure
* other primary anxiety disorder and major psychosis
* use hormone therapy
* use herb medicine

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale | 4 weeks aftter ear acupressure

SECONDARY OUTCOMES:
Menopause Rating Scale,Short Form Health Survey(SF-36),CGI | 4 weeks aftter ear acupressure

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Ling Kao, MD, Principal Investigator — Chang-Hua Hospital, Department of Health
Locations (1):
- Chang-Hua Hospital, Changhua, Taiwan